CLINICAL TRIAL: NCT03919435
Title: Trimethoprim-Sulfamethoxazole Effects on the Nasal Microbiome in Granulomatosis With Polyangiitis
Brief Title: TEMPO Study: Trimethoprim-Sulfamethoxazole in Granulomatosis With Polyangiitis
Acronym: TEMPO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Rennie Rhee, M.D., MSCE, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 831864
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Granulomatosis With Polyangiitis; Wegener Granulomatosis
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- On Drug (Experimental)
  Interventions: Drug: Trimethoprim Sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim Sulfamethoxazole — Dosage: 160mg-800mg Frequency: 2 times a day Dosage Form: Pill (oral) Duration: 4 weeks

SUMMARY:
Granulomatosis with polyangiitis (GPA; Wegener's) is a multi-organ autoimmune disease characterized by necrotizing granulomatous inflammation and vasculitis. Upper respiratory involvement occurs in up to 90% of patients with GPA and is often the first manifestation of the disease. Patients with upper respiratory tract disease are more at risk of local and systemic relapse. Microbial organisms may be involved in inducing disease activity in GPA. Previous culture-dependent studies found that patients with GPA were more likely to be chronic nasal carriers of Staphylococcus aureus compared to non-GPA chronic rhinosinusitis and healthy controls; additionally, GPA patients with S. aureus colonization are more likely to experience a future relapse. This led to a randomized placebo-controlled trial of trimethoprim-sulfamethoxazole (TMP-SMX) which showed this antibiotic/antifungal was effective in preventing relapse in GPA. Whether the benefits of TMP-SMX are related to its antimicrobial properties versus anti-inflammatory effects is still unknown. The objective of this study is to prospectively evaluate the changes in the nasal microbiome, mycobiome, and host immunity in patients with GPA before, during, and after receipt of TMP-SMX for 4 weeks. The target enrollment number is 30 participants, and the investigators will include patients seen at the Penn Vasculitis Center with GPA (diagnosed according to the American College of Rheumatology Classification Criteria or based on investigator's judgment). To analyze nasal microbiome and host immunity, participants will be swabbed with nasal swab and cytobrush for DNA sequencing and other studies. An optional research blood draw is also included. The investigators and coordinators will follow each patient longitudinally over a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 year of age or older
* Both male and female gender will be included
* Patients with GPA will be defined according to classification criteria or according to the investigator's judgment
* Patients must have history of sinonasal involvement related to GPA
* Patients must also be in remission for at least 3 months and expect to remain on stable immunosuppressive therapies for the next 24 weeks, with the exception of minor prednisone changes
* Prednisone dose or equivalent less than or equal to 10mg at enrollment

Exclusion Criteria:

* Receipt of oral antibiotics or antifungals within past 6 weeks including antimicrobials for prevention of Pneumocystis jiroveci pneumonia
* Infection involving sinuses or nose in past 4 weeks
* Receipt of topical nasal antibiotics (including mupirocin) within the past 4 weeks
* Contra-indication or prior adverse reaction to TMP-SMX such as sulfa allergy, severe renal insufficiency (CrCl < 15 ml/min) or severe hepatic failure according to most recent labs in past 6 months
* At risk for drug interactions related to TMP-SMX
* Intra-nasal cocaine use in prior 3 months
* Known history of HIV or primary immunodeficiency syndrome
* Pregnant or planning to become pregnant in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
nasal microbiome in relative abundance ( host gene expression in proportion) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States